CLINICAL TRIAL: NCT06914713
Title: Efficacy Evaluation of Jin-shui Huan-xian Formula in Retarding the Decline of Pulmonary Function in IPF
Brief Title: Jin-shui Huan-xian Formula for Retarding the Decline of Pulmonary Function in IPF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM for IPF
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Pulmonary Fibrosis(IPF)
Keywords: Idiopathic Pulmonary Fibrosis; traditional Chinese medicine; randomized controlled trial; pulmonary function
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jin-shui Huan-xian granule in addition to the guideline - directed treatment. (Experimental): The experimental group was given Jin-shui Huan-xian Formula in addition to the treatment guided by the guideline "Idiopathic Pulmonary Fibrosis (an Update) and Progressive Pulmonary Fibrosis in Adults: An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline ".
  Interventions: Drug: Jin-shui Huan-xian granule
- Jin-shui Huan-xian granule placebo in addition to the guideline - directed treatment. (Placebo Comparator): The experimental group was given Jin-shui Huan-xian granule placebo in addition to the treatment guided by the guideline"Idiopathic Pulmonary Fibrosis (an Update) and Progressive Pulmonary Fibrosis in Adults: An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline ".
  Interventions: Drug: Jin-shui Huan-xian granule placebo

INTERVENTIONS:
Drug: Jin-shui Huan-xian granule — Jin-shui Huan-xian Granules: on the basis of treatment guided by "Idiopathic Pulmonary Fibrosis (an Update) and Progressive Pulmonary Fibrosis in Adults: An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline ", the experimental group was given Jin-shui Huan-xian Granules for treatment. The granules were taken orally, 1 dose per day, twice a day, and the continuous administration lasted for 52 weeks.
  Other Names: Jin-shui Huan-xian Granules
  Arms: Jin-shui Huan-xian granule in addition to the guideline - directed treatment.
Drug: Jin-shui Huan-xian granule placebo — Jin-shui Huan-xian granule placebo: on the basis of treatment guided by "Idiopathic Pulmonary Fibrosis (an Update) and Progressive Pulmonary Fibrosis in Adults: An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline ", the experimental group was given Jin-shui Huan-xian Granules placebo for treatment. The granules were taken orally, 1 dose per day, twice a day, and the continuous administration lasted for 52 weeks.The Jin-shui Huan-xian granules and their placebo are identical in appearance, weight, color and smell.
  Arms: Jin-shui Huan-xian granule placebo in addition to the guideline - directed treatment.

SUMMARY:
This study is to evaluate the clinical efficacy and safety of Jin-shui Huan-xian Formula in retarding the decline of pulmonary function in IPF, generate high - quality clinical evidence, and establish a treatment plan of Jin-shui Huan-xian Formula for retarding the decline of pulmonary function in Idiopathic Pulmonary Fibrosis（IPF）

DETAILED DESCRIPTION:
The study took 384 IPF patients as the research objects and adopted a randomized, double - blind, placebo - controlled trial design. The patients were randomly divided into an experimental group and a control group. On the basis of guideline - guided treatment, the experimental group was given Jin-shui Huan-xian Formula, and the control group was given a placebo of Jin-shui Huan-xian Formula. The treatment lasted for 52 weeks. Pulmonary function (FVC) was set as the primary outcome indicator, and acute exacerbation, pulmonary function (DLCO, DLCO%, etc.), exercise endurance, quality of life, etc. were set as secondary outcome indicators. Blood routine, urine routine, liver function, renal function, electrocardiogram, etc. were set as safety indicators. The clinical efficacy and safety of Jin-shui Huan-xian Formula in retarding the decline of pulmonary function in IPF were evaluated to generate high - quality clinical evidence and establish a treatment plan of Jin-shui Huan-xian Formula for retarding the decline of pulmonary function in IPF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria for IPF.
2. Pulmonary function: The percentage of forced vital capacity (FVC) to the predicted value is ≥ 50%; and the percentage of the diffusing capacity of the lung for carbon monoxide (DLCO) to the predicted value is ≥ 30%.
3. Patients who meet the syndrome - differentiation criteria for lung - qi deficiency syndrome, lung - and - kidney qi deficiency syndrome, etc.
4. Aged between 40 and 85 years old.
5. Patients who voluntarily accept the treatment and sign the informed consent

Exclusion Criteria:

1. Patients in the acute exacerbation phase of IPF.
2. Patients complicated with other pulmonary diseases such as chronic obstructive pulmonary disease (COPD), lung cancer, active pulmonary tuberculosis, bronchiectasis, and pulmonary embolism.
3. Patients with severe joint, peripheral nerve, and peripheral vascular diseases that affect limb movement and who are bed - ridden for a long time and cannot complete the six - minute walk test.
4. Patients complicated with severe cardiovascular and cerebrovascular diseases (malignant arrhythmia, unstable angina pectoris, acute myocardial infarction, heart function grade 3 or above, stroke, cerebral hemorrhage, etc.).
5. Patients complicated with liver diseases such as cirrhosis or secondary portal hypertension, bleeding caused by esophageal and gastric varices, patients with kidney diseases requiring dialysis or kidney transplantation, or patients with abnormal liver and kidney functions (ALT, AST, and BUN are 1.5 times higher than the upper limit of the normal range, and blood Cr is higher than the upper limit of the normal range).
6. Patients with unclear consciousness, various mental illnesses, etc., who cannot communicate normally.
7. Pregnant or lactating women and patients with a recent plan for pregnancy.
8. Patients who have participated in other clinical trials within 1 month before enrollment.
9. Patients known to be allergic to any of the test medications and their components.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | The change in absolute FVC value before treatment and at 52 weeks of treatment
  FVC will be used to assess pulmonary function.

SECONDARY OUTCOMES:
The time of the first acute exacerbation | Up to week 52.
  The time of the patients' first acute exacerbation will be recorded.
Frequency of acute exacerbation | Up to week 52
  Frequency of acute exacerbation will be recorded.
Frequency of acute exacerbations resulting in hospitalization | Up to week 52
  Frequency of acute exacerbation resulting in hospitalization will be recorded.
Frequency of acute exacerbations resulting in ICU admission | Up to week 52
  Frequency of acute exacerbation resulting in ICU admission will be recorded.
Annual acute exacerbation rate | Up to week 52
  The annual acute exacerbation rate will be calculated in each group at the end of the trial.
Annual hospitalization rate due to acute exacerbation | Up to week 52
  The Annual hospitalization rate due to acute exacerbation will be calculated in each group at the end of the trial.
Annual rate of ICU admission due to acute exacerbation | Up to week 52.
  The Annual ICU admission rate due to acute exacerbation will be calculated in each group at the end of the trial.
Diffusing Capacity of Carbon Monoxide（DLCO） | Change from baseline DLCO at week 13, 26, 39 and 52.
  DLCO will be used to assess pulmonary function.
Percent of Diffusing Capacity of Carbon Monoxide（DLCO%） | Change from baseline DLCO% at week 13, 26, 39 and 52.
  DLCO% will be used to assess pulmonary function.
Percent of Forced Vital Capacity（FVC%） | Change from baseline FVC%at week 13, 26, 39 and 52.
  FVC% will be used to assess pulmonary function.
Alveolar ventilation（VA） | Change from baseline VA at week 13, 26, 39 and 52.
  VA will be used to assess pulmonary function.
.Diffusion capacity for carbon monoxide per liter of alveolar volume（DLCO/VA） | Change from baseline DLCO/VA at week 13, 26, 39 and 52.
  DLCO/VA will be used to assess pulmonary function.
All-cause mortality rate | Up to week 52.
  The all-cause mortality rate will be calculated in each group at the end of the trial.
Mortality rate due to acute exacerbation | Up to week 52.
  The mortality rate due to acute exacerbation will be calculated in each group at the end of the trial.
Progression-Free Survival（PFS） | Up to week 13, 26, 39 and 52.
  According to "Idiopathic Pulmonary Fibrosis in Adults (Update) and Progressive Pulmonary Fibrosis: An Official Clinical Practice Guideline of the ATS/ERS/JRS/ALAT ": The time from enrollment to the first meeting of disease progression (at least two of respiratory symptoms, physiological evidence and radiological evidence).
Six Minute Walk Test (6MWT) | Change from baseline 6MWT at week 13, 26, 39 and 52.
  6MWT will be applied to evaluate the exercise capacity. The higher values indicate the better exercise capacity.
Imaging findings | Up to week 26, 52.
  Changes in chest CT imaging will be assessed before and after JSHX treatment to evaluate its impact on pulmonary fibrosis in IPF patients. High-resolution computed tomography (HRCT) will be used to quantify alterations in lung parenchyma, including ground-glass opacities, reticulation, and honeycombing. Quantitative software-based analysis (e.g., histogram-based texture analysis) may be applied to standardize the evaluation. Radiologists blinded to treatment allocation will independently review the images to ensure objectivity.
A Tool to Assess Quality of life (ATAQ-IPF) | Change from baseline ATAQ-IPF scores at week 13, 26, 39 and 52.
  ATAQ - IPF is currently a specialized scale for evaluating the quality of life of patients, consisting of 13 dimensions and 74 items, with each item being scored from 1 to 5 points. A higher score indicates a worse condition.
Idiopathic pulmonary fibrosis patient reported outcomes (IPF-PRO) | Change from baseline SGRQ scores at week 13, 26, 39 and 52.
  IPF-PRO is a scale used to evaluate the quality of life of patients, where patients recall their condition over the past two weeks based on their subjective experience. The evaluation covers four domains: Physiological, Psychological, Environmental, and Satisfaction, comprising 18 items in total. Higher scores indicate worse conditions.
Dyspnea | Change from baseline CAT scores at week 13, 26, 39 and 52.
  Dyspnea will be assessed by 22.modified Medical Research Council(mMRC) scores. A score of 0-4 will be given according to the degree of immediate dyspnea. A higher score indicates a worse condition.
Cough Visual analog scale(VAS) | Change from baseline CAT scores at week 13, 26, 39 and 52.
  The Cough VAS is a method of quantitatively assessing cough symptoms using the Visual Analogue Scale. The score ranges from 1 to 100, a higher score indicates a worse condition.
Clinical symptoms and Signs | Change from baseline clinical symptoms and signs up at week 13, 26, 39 and 52.
  Clinical symptoms and Signs will be evaluated through a scale. The scale includes coughing, expectoration, chest tightness, shortness of breath, wheezin. The Clinical Symptom Rating Scale includes 6 items: cough, expectoration, chest tightness, shortness of breath, wheezing, and cyanosis. Each item has a score of 0-3, totaling 18 points. The higher the score, the worse he patient's condition.
Krebs Von den Lungen-6 (KL-6) | Change from baseline KL-6 level at week 13, 26, 39 and 52.
  Detect the level of KL-6.
Interleukin-6 (IL-6) | Change from baseline IL-6 level at week 13, 26, 39 and 52.
  Detect the level of IL-6.
Ferritin | Change from baseline Ferritin level at week 13, 26, 39 and 52.
  Detect the level of Ferritin.
Immunoglobulin | Change from baseline immunoglobulins level at week 13, 26, 39 and 52.
  Detect the level of immunoglobulins
T, B and NK lymphocyte subsets | Change from baseline T, B and NK lymphocyte subsets level at week 13, 26, 39 and 52.
  Detect the level of T, B and NK lymphocyte subsets. The common indicators of TBNK lymphocyte subsets and their respective units of measurement are as follows: the total T cells (CD3+), measured in cells per microliter (cells/µL); the helper T cells (CD3+CD4+), measured in cells/µL; the cytotoxic T cells (CD3+CD8+), measured in cells/µL; the B cells (CD19+), measured in cells/µL; the natural killer cells (NK cells, CD16+CD56+, CD3-), measured in cells/µL; and the CD4/CD8 ratio, which is a unitless ratio. These indicators are detected by flow cytometry and can reflect the immune function status of the body.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan, China